CLINICAL TRIAL: NCT02831660
Title: A Compassionate Use Program of Idarucizumab for Reversal of the Anticoagulant Effects of Dabigatran in Japanese Patients Who Have Uncontrolled Bleeding or Require Emergency Surgery or Procedures
Brief Title: CU Programme of Idarucizumab for Japanese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1321.14
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

ARMS (1):
- idarucizumab (Experimental)
  Interventions: Drug: idarucizumab

INTERVENTIONS:
Drug: idarucizumab

SUMMARY:
The objective is to collect the safety data of idarucizumab for patients treated with dabigatran who require rapid reversal of the anticoagulant effects of dabigatran in cases of uncontrolled or life-threatening bleeding or when emergency surgery or urgent procedures are required.

ELIGIBILITY:
Inclusion criteria:

* Currently taking dabigatran etexilate.
* Age >= 20 years at entry.
* Written Informed consent
* Group A:

  -- Uncontrolled or life-threatening judged by the physician to require a reversal agent.
* Group B:

  * A condition requiring emergency surgery or invasive procedure where adequate hemostasis is required. Emergency is defined as within the following 8 hours.

Exclusion criteria:

* Contraindications to study medication including known hypersensitivity to the drug or its excipients (subjects with hereditary fructose intolerance may react to sorbitol).
* Group A:

  * Patients with minor bleeding (e.g. epistaxis, hematuria) who can be managed with standard supportive care.
  * Patients with no clinical signs of bleeding.
* Group B:

  * surgery or procedure which is elective or where the risk of uncontrolled or unmanageable bleeding is low.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Fukuoka Tokushukai Medical Center, Fukuoka, Kasuga, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Idarucizumab 5 g: The total dose of 5 g (two 2.5 g vials) was administered intravenously. A single vial contained 2.5 g of idarucizumab (in buffered solution for injection). Patients received a 2.5 g vial of study medication and a second 2.5 g vial within the next 15 minutes. In rare instances, an additional 5 g dose was to be justified.
Period: Overall Study
Arm/Group | Idarucizumab 5 g
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) comprised all patients who had been received at least 1 dose of the study medication.
Arm/Group | Idarucizumab 5 g
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug-related adverse events is presented
Time Frame: from first drug administration until 5 days after last drug administration, up to 6 days.
Population: Treated Set
Measure: Number; unit: Percentage of participants
Arm/Group | Idarucizumab 5 g
Number analyzed (Participants) | 1
Percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 5 days after last drug administration, up to 6 days.
Arm/Group | Idarucizumab 5 g
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idarucizumab 5 g (N=1)
Platelet count decreased (Investigations) | 1

LIMITATIONS AND CAVEATS:
Because of the trial design and backgrounds, only 1 patient was entered in the trial. Because of the limited number of patients, it was difficult to draw general conclusion regarding safety or tolerability of idarucizumab

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.